CLINICAL TRIAL: NCT01941056
Title: Phase I Evaluation of a CMV-MVA Triplex Vaccine: Safety and Biologically Effective Dose in Healthy Volunteers With or Without Prior Immunity to CMV and Vaccinia
Brief Title: Vaccine Therapy in Healthy Volunteers With or Without Previous Exposure to Cytomegalovirus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 08173; NCI-2013-01625 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 08173 (Other: City of Hope Medical Center); R01CA077544 (NIH)
Record Dates: First submitted 2013-09-05; First posted 2013-09-13 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Cytomegalovirus Infection; Healthy, no Evidence of Disease
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (CMV-MVA Triplex vaccine) (Experimental): Participants receive multi-CMV epitope modified vaccinia Ankara vaccine IM followed by a booster injection 28 days later in the absence of unacceptable toxicity.
  Interventions: Biological: multi-CMV epitope modified vaccinia Ankara vaccine; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: multi-CMV epitope modified vaccinia Ankara vaccine — Given IM
  Other Names: CMV-MVA triplex vaccine
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and the best dose of vaccine therapy in healthy volunteers with or without previous exposure to cytomegalovirus. Vaccines made from a gene-modified virus may help the body build an immune response and may help prevent cytomegalovirus infection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish a biological optimal dose of the cytomegalovirus (CMV)-modified vaccinia Ankara (MVA) Triplex vaccine (multi-CMV epitope modified vaccinia Ankara vaccine).

II. To determine if the vaccine is safe and well tolerated in healthy volunteers at these doses.

SECONDARY OBJECTIVES:

I. To provide preliminary evidence of CMV-MVA Triplex vaccine driven expansion of CMV-specific immune responses that would support further evaluation of this vaccine in hematopoietic cell transplantation (HCT) recipients.

II. To confer CMV-specific immunity to CMV-negative volunteers and to determine the duration of immune enhancement of CMV-specific cell mediated immunity (CMI) function up to 12 months following immunization of healthy volunteers.

OUTLINE: This is a dose-escalation study.

Participants receive multi-CMV epitope modified vaccinia Ankara vaccine intramuscularly (IM) followed by a booster injection 28 days later in the absence of unacceptable toxicity.

After completion of study treatment, participants are followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Sodium range from within normal institutional limits to less than a grade I toxicity
* Potassium range from within normal institutional limits to less than a grade I toxicity
* Chloride range from within normal institutional limits to less than a grade I toxicity
* Carbon dioxide range from within normal institutional limits to less than a grade I toxicity
* Glucose range from within normal institutional limits to less than a grade I toxicity
* Alkaline phosphatase (AP) range from within normal institutional limits to less than a grade I toxicity
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) range from within normal institutional limits to less than a grade I toxicity
* Blood urea nitrogen (BUN) range from within normal institutional limits to less than a grade I toxicity
* Creatinine range from within normal institutional limits to less than a grade I toxicity
* Lactic dehydrogenase (LDH) range from within normal institutional limits to less than a grade I toxicity
* Total bilirubin range from within normal institutional limits to less than a grade I toxicity
* Uric acid range from within normal institutional limits to less than a grade I toxicity
* Albumin > lower limit of normal institutional limits
* White blood count range from within normal institutional limits to less than a grade I toxicity
* Hemoglobin (HGB) range from within normal institutional limits to less than a grade I toxicity
* Hematocrit (HCT) range from within normal institutional limits to less than a grade I toxicity
* Platelet count is within the lower limit of normal institutional limits and not more than 1.5 times the upper limit of normal institutional limits
* Hepatitis B virus (HBV) surface antigen negative and hepatitis C virus (HCV) seronegative; human immunodeficiency virus (HIV)-1 seronegative
* Currently not taking daily medications for chronic or intercurrent illness; those medications which are excepted from this rule are thyroid replacement, estrogen replacement, dietary vitamins and protein supplements, and any medications not known or likely to be immunosuppressive, as determined by the principal investigator (PI)
* No surgery in past 6 months which required general anesthesia, but minor procedures, such as dental surgery and superficial diagnostic biopsies, are permitted
* No diagnosis which has been associated with immunodeficiency
* No active infection for which the subject is receiving treatment
* Framingham Risk Score for cardiovascular disease =< 10%; no history of heart disease, e.g. previous treated arrhythmia or myocardial infarction; no horizontal positioning-induced or activities of normal living exercise-induced shortness of breath; no history of stroke or claudication; no current treatment with medication for high cholesterol or other lipid abnormality; a documented electrocardiogram (ECG) and cardiac troponin must be within normal institutional limits in the past 30 days; "normal ECG with sinus tachycardia" or " normal ECG with sinus bradycardia" is allowable based on a history of absent cardiac/exercise related symptoms as determined by the P.I. in consultation with a senior staff cardiologist
* No history of or prior treatment for diabetes type 1 or diabetes type 2
* Women of childbearing age must have a negative urine pregnancy test and must not be planning to become pregnant within the next 6 months
* No history of adverse events with a prior smallpox vaccination

SECONDARY ELIGIBILITY CRITERIA:

* It is anticipated that there could be a delay of 1-3 months between screening and actual vaccination; alternatively, there could be a delay due to availability of the vaccine; therefore, prior to registration for vaccination, the following secondary eligibility criteria must be met:
* If not tested in past 4 months, serum chemistries and blood counts are within normal limits; hepatitis B virus (HBV) surface antigen negative and hepatitis C virus (HCV) seronegative; HIV-1 antibody negative
* Women of childbearing age must have a urine pregnancy test performed within 48 hours of each vaccine administration with a negative result
* Laboratory values prior to booster injection may include grade 1 laboratory abnormalities, but any grade >= grade 2 will exclude the subject from a booster injection

Exclusion Criteria:

* Any previous condition, or one that becomes known during the screening period, that would suggest that the individual could be immunologically impaired, or for which this study would pose a danger to him/herself or about which the P.I., in evaluating the subject for eligibility, determines that this exclusion is appropriate
* Subjects are excluded who have a history of cancer other than basal cell skin cancer, or any condition, psychiatric or otherwise, that would preclude informed consent, consistent follow-up or compliance with any aspect of the study (e.g., untreated schizophrenia or other significant cognitive impairment, etc. as determined by the PI. In addition, allergic diatheses as define by a history of asthma, anaphylaxis, or generalized urticaria, or by daily use of antihistamines, episodic (more than once in past 3 months) inhalational medications including steroidal agents, non-steroidal agents, or cromolyn sodium
* Subjects with severe migraine headaches (more than one per month on average in the past 6 months or requiring preventive medications) are excluded
* Any of the following cardiac findings of ECG abnormality:

  * Conduction disturbance (complete left or right bundle branch block, intraventricular conduction disturbance with QRS > 120 ms, atrioventricular block [AV] block of any degree, and corrected QT [QTc] prolongation > 450 msec for men and > 460 msec for women)
  * Repolarization (ST segment or T wave) abnormality
  * Significant atrial or ventricular arrhythmia, including frequent ectopy (e.g., 2 premature ventricular contractions in a row; and
  * Evidence of past myocardial infarction
* Any previous condition, or one that becomes known during the screening period, that would suggest that the technicians and health professionals involved in the study would be exposed to specific infectious risk
* Treatment with whole or subunit CMV or poxvirus vaccine in the last 12 months
* Men with partners of child-bearing potential and women of child-bearing potential who are not willing to use medically effective birth control methods, e.g. contraceptive pill, condom, or diaphragm, and continue this for 6 weeks after the second and last dose of vaccine
* Subjects who have had a live vaccine =< 30 days prior to administration of study vaccine or subjects who are =< 2 weeks within administration of inactivated vaccines (e.g. influenza vaccine)
* Persons who are employed by or are a student at City of Hope and are in a chain of command that reports directly to persons listed on the protocol as Principal Investigator or Co-Investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01-05 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2017-07-28 (Actual)

PRIMARY OUTCOMES:
Successful completion of 2 injections without dose-limiting toxicity (DLT) according to the Division of Microbiology and Infectious Diseases (DMID) adult toxicity tables | Up to 28 days

SECONDARY OUTCOMES:
Evidence of CMV-MVA Triplex vaccine driven expansion of CMV-specific immune responses to support further evaluation of this vaccine in HCT recipients. | Up to 1 year
  Expansion of CMV-specific T-cells in peripheral blood mononuclear cell (PBMC)will be evaluated by flow cytometry, immunocytochemistry (ICC) assays, and enzyme-linked immunosorbent spot (ELISPOT)
Frequency of polyfunctional cluster of differentiation (CD)4+ and CD8+ T cells recognizing CMV Ag, expressed as concentrations | Up to 1 year
  A one-sample signed-rank test will be used to compare pre- and post-vaccination CD4+ and CD8+ T cell levels. A secondary analysis will model cell concentrations as a function of time, dose, and CMV serostatus. Mixed models and generalized estimating equations will be used to permit quantitative estimation and flexible investigation of potentially interacting covariables.

CONTACTS AND LOCATIONS:
Overall Officials: John Zaia, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States